CLINICAL TRIAL: NCT03311347
Title: Influence of Hyperoxia and Hypobaria on Atelectasis Occurrence and Mitigation of Atelectasis Formation
Brief Title: Atelectasis Formation: Role of Positive Pressure Breathing, Hyperoxia, and Hypobaria
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Direction Centrale du Service de Santé des Armées (Other)
Collaborators: Uppsala University Hospital (Other); Percy Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: PDH1-SMO2-0714
Record Dates: First submitted 2017-04-05; First posted 2017-10-17 (Actual); Last update posted 2019-05-14 (Actual); Status verified 2019-05

CONDITIONS: Pulmonary Atelectasis
Keywords: pulmonary ultrasound; hypergravity; human physiology; oxygen; lung ventilation; lung perfusion; computed tomography; electrical impedance tomography; altitude chamber
MeSH Terms: conditions — Pulmonary Atelectasis | interventions — Intermittent Positive-Pressure Ventilation

STUDY DESIGN:
Intervention Model Description: Two arms are studied, breathing air or 100%O2. In each arm, subjects are studied at two occasions: with and without positive pressure breathing. These occasions are randomized.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 100%O2 breathing (Experimental): Primary aim, item 1
  Interventions: Other: +Gz accelerations and positive pressure breathing
- Air breathing (Experimental): Primary aim, item 1
  Interventions: Other: +Gz accelerations and positive pressure breathing

INTERVENTIONS:
Other: +Gz accelerations and positive pressure breathing

SUMMARY:
The primary aim of this project is to get further knowledge of the physiology of flight atelectasis and its prevention. We seek to: 1) assess whether low levels of positive pressure breathing can prevent atelectasis formation in humans during exposure to hyperoxia and +Gz-accelerations. 2) get further knowledge on the effects of hypobaria on regional ventilation and perfusion.

A secondary aim is to evaluate the effect of anti G-trouser inflation on ventilation and regional perfusion.

DETAILED DESCRIPTION:
The effect of positive pressure breathing on lung function is being studied, when applied during exposure to hyperoxia and +Gz-accelerations. Focus is on lung tissue compression, ventilation and regional perfusion. In addition, the influence of hypobaria on these parameters is assessed.

This study is conducted in accordance with the amended Declaration of Helsinki. The Ethics Committee Ile-de-France III (ref. 3274) and the French National Agency for Drug Safety ANSM have approved the protocol (ref. ID RCB 2015-A00485-44 and ANSM 151046B-32).

Primary aim, item 1: Experiments are conducted in a human centrifuge. The protocol mimics a routine peacetime flight in combat aircraft, and includes 1hr05 min at +1Gz followed by 10-min exposure to +1.4 to +3.5Gz . Subjects are exposed three times to this sequence, breathing at positive pressure levels of 0, 5 or 10 hPa. Two groups of sixteen healthy male non-smoking volunteers, wearing anti-G trousers, are studied and compared: group 1 breathes air, group 2 100% O2.

Primary aim, item 2: Experiments are conducted in a hypobaric chamber. Sixteen healthy male non-smoking volunteers are exposed to four conditions: 0 or 15,000 ft altitude, breathing air or 100%O2. Protocol duration is 1h15min. Positive breathing pressure can be applied depending on the results of the experiments of item 1.

Secondary aim: Experiments are conducted in a human centrifuge. Sixteen healthy male non-smoking volunteers are exposed to four conditions: uninflated or inflated anti-G trousers (175 hPa), +1 or +3.5 Gz for 3 min.

ELIGIBILITY:
Inclusion Criteria:

* normal lung function checked by pulmonary function tests.
* normal ECG
* normal clinical examination

Aim 1 exclusion criteria:

* smoking
* myopia
* past medical history of heart or lung disease
* current medical treatment for heart or lung disease
* past medical history of back pain or spine trauma or disease
* otitis
* bad tolerance to +Gz accelerations (G-induced loss of consciousness, motion sickness)
* claustrophobia in the centrifuge gondola

Aim 2 exclusion criteria:

* smoking
* past medical history of heart or lung disease
* current medical treatment for heart or lung disease
* otitis
* bad tolerance to the altitude chamber (15,000 ft): ear pain, claustrophobia

Ages: 25 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2015-09-14 (Actual); Primary Completion 2019-06-30 (Estimated); Study Completion 2020-01-01 (Estimated)

PRIMARY OUTCOMES:
atelectasis formation (change between pre and post-protocol) | pre-protocol (baseline) and 1h30 min after centrifuge stop
  computerized tomography: 0-5 scale for size and localization
change in pulmonary ventilation between 1 Gz, 1.6 Gz and 3.5 Gz | pre-protocol (baseline), baseline + 1hr, baseline +1h10 min, baseline +1h15 min
  electrical impedance tomography: deltaZ on regions of interest
change in pulmonary tissue density from baseline at centrifuge stop and 1h30 min after stop | pre protocol (baseline), at centrifuge stop (baseline + 1h15 min) and 1h30 min after centrifuge stop
  ultrasound: number of lung comets + localization

CONTACTS AND LOCATIONS:
Overall Officials: Dominique Felten, MD, Study Chair — Armed Forces Biomedical Research Institute
Locations (2):
- France (2):
  - Armed Forces Biomedical Research Institute, Brétigny-sur-Orge
  - Department of Radiology, Percy hospital, Clamart

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dussault C, Gontier E, Verret C, Soret M, Boussuges A, Hedenstierna G, Montmerle-Borgdorff S. Hyperoxia and hypergravity are independent risk factors of atelectasis in healthy sitting humans: a pulmonary ultrasound and SPECT/CT study. J Appl Physiol (1985). 2016 Jul 1;121(1):66-77. doi: 10.1152/japplphysiol.00085.2016. Epub 2016 Apr 21. PMID 27103651
- [Result] Borges JB, Hedenstierna G, Bergman JS, Amato MB, Avenel J, Montmerle-Borgdorff S. First-time imaging of effects of inspired oxygen concentration on regional lung volumes and breathing pattern during hypergravity. Eur J Appl Physiol. 2015 Feb;115(2):353-63. doi: 10.1007/s00421-014-3020-9. Epub 2014 Oct 17. PMID 25323531